CLINICAL TRIAL: NCT02233439
Title: Efficacy of Herbal Galactogogues: a Double-blinded, Placebo-controlled Randomized Trial.
Brief Title: Double-blind, Placebocontrolled A Randomized Trial on the Efficacy of Herbal Galactogogues
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Collaborators: Milte Italia SpA (Unknown)
Responsible Party: Principal Investigator, Antonella Cromi, Associate professor, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 54/2013
Record Dates: First submitted 2014-08-29; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Breastfeeding
Keywords: galactagogues; herbs; breastfeeding; supplements; Silybum marianum; Galega officinalis
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): a placebo identical in appearance to the galactagogue product
  Interventions: Dietary Supplement: Placebo
- No treatment (No Intervention): Usual care and breastfeeding support
- Herbal galactagogue (Experimental): A commercially available product containing a combination of Silybum marianum 400 mg and Galega officinalis 150 mg, once a day for 6 weeks
  Interventions: Dietary Supplement: Herbal galactagogue

INTERVENTIONS:
Dietary Supplement: Herbal galactagogue
  Other Names: Piùlatte® Plus (MILTE ITALIA SpA)
  Arms: Herbal galactagogue
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness of a commercially available product containing a combination of Silybum marianum and Galega officinalis to support continuation or augmentation of breast milk production.

ELIGIBILITY:
Inclusion Criteria:

* singleton, term delivery
* >2.5 kg newborn weight
* lactation-deficiency

Exclusion Criteria:

* Neonatal Intensive Care Unit admission
* use of galactagogue drugs
* allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-01 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of mothers who exclusively breastfeed their child | At 6 weeks postpartum

SECONDARY OUTCOMES:
Rate of breastfeeding (either exclusively or as a supplement to formula feeding ) | at 6 weeks and 3 months
Volume (mL) and frequency (times a day) of formula | 6 weeks postpartum
weight gain experienced by the newborns | 6 weeks postpartum
serum prolactin level | at baseline and 6 weeks after treatment
Rate of maternal allergic reactions and gastrointestinal side effects | 6 weeks postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria Ospedale di Circolo e Fondazione Macchi, Presidio F. Del Ponte, Varese, Italy

REFERENCES:
- [Derived] Foong SC, Tan ML, Foong WC, Marasco LA, Ho JJ, Ong JH. Oral galactagogues (natural therapies or drugs) for increasing breast milk production in mothers of non-hospitalised term infants. Cochrane Database Syst Rev. 2020 May 18;5(5):CD011505. doi: 10.1002/14651858.CD011505.pub2. PMID 32421208